CLINICAL TRIAL: NCT01469780
Title: Assessing Pain as a Mediator of Behavior Change in Post-coronary Angioplasty Patients
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 9806003392; 3P30AG022845-07S1 (NIH)
Record Dates: First submitted 2011-11-08; First posted 2011-11-10 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Pain; Depressive Symptoms; Quality of Life
Keywords: Pain; Health behavior change; Coronary angioplasty; Cardiovascular disease; Outcomes; Morbidity; Mortality
MeSH Terms: conditions — Pain; Depression; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The focus of this secondary data analysis is to determine whether pain due to a combination of both cardiac and non cardiac sources operates as a mediator of behavior change, an area that has not been previously evaluated.

DETAILED DESCRIPTION:
This is a secondary data analysis of an existing dataset generated from The Healthy Behavior Trial, an NHLBI-funded randomized controlled trial that enrolled 660 post-coronary angioplasty patients between October 1999 and March 2001. This study employed a behavioral intervention to motivate PCI patients to adopt health behaviors in order to reduce major cardiac and neurologic morbidity and mortality. Patients in the experimental arm were told their estimated biologic age (calculated from the health risk assessment) and risk factors were presented in terms of "biologic age reduction" that could be achieved if a change was made in each health behavior area. Those in the control arm were provided with risk factors (also obtained from the health risk assessment) and told that changing each health behavior could "increase your lifespan."

Specific Aims:

Utilizing 12 month longitudinal data for patients with cardiovascular disease who have undergone coronary angioplasty we will:

Specific aim 1: Determine if pain is a mediator of health behavior change over 12 months.

Specific aim 2: Assess behavior change patterns over 12 months, stratifying for degree of pain, depression and/or stress.

Specific aim 3: Evaluate the effect of pain on quality of life (physical, social, role-physical, role-emotional, vitality, mental health, bodily pain and general health domains), combined major cardiac and neurologic morbidity/mortality and hospitalizations over 12 months.

ELIGIBILITY:
Inclusion Criteria:

* all patients in the database who had participated in the Healthy Behavior Trial. The Healthy Behavior Trial was a randomized controlled trial of a psychoeducational intervention designed to motivate multi-behavior change (changing 2 or more cardiovascular risk factors) in post-coronary angioplasty patients over the course of 24 months.

Exclusion Criteria:

* Non-participants in the Healthy Behavior Trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The is a database study of a cohort of 660 patients with cardiovascular disease who had recently undergone coronary angioplasty.
Sampling Method: Probability Sample
Enrollment: 660 (Actual)
Dates: Start 1999-04; Primary Completion 2003-08 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
successful behavior change over 12 months | Baseline, 3, 6, 9 and 12 months
  Health behavior will be examined in five areas: overall physical activity, strength training, aerobic activity, weight loss, and smoking cessation. Successful health behavior change will be defined as "action" (engaging in the behavior < six months) or "maintenance" (engaging in the behavior ≥ six months to five years), according to the Transtheoretical Model. We will use self-reported data.

SECONDARY OUTCOMES:
Quality of life | Within-patient change from baseline to 12 months
  The SF-36 health survey will be the primary measure of quality of life. Each of the eight individual domain scores will be evaluated (physical, social, role-physical, role-emotional, vitality, mental health, bodily pain and general health) and the within-patient change from baseline to 12 months will be calculated. The physical and mental component summary measures will also be calculated, as will the within-patient change from baseline to 12 months for the component scores. We will assess these measures as both continuous and dichotomous measures.

CONTACTS AND LOCATIONS:
Overall Officials: Janey C Peterson, EdD, MS, RN, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

REFERENCES:
- [Background] Charlson ME, Peterson JC, Boutin-Foster C, Briggs WM, Ogedegbe GG, McCulloch CE, Hollenberg J, Wong C, Allegrante JP. Changing health behaviors to improve health outcomes after angioplasty: a randomized trial of net present value versus future value risk communication. Health Educ Res. 2008 Oct;23(5):826-39. doi: 10.1093/her/cym068. Epub 2007 Nov 19. PMID 18025064
- See also: Related Info — http://tripll.org/